CLINICAL TRIAL: NCT05955417
Title: The Development and Validation of a Novel Equation for Estimating Sodium Intake in Peritoneal Dialysis
Brief Title: A Novel Equation for Estimating Sodium Intake in Peritoneal Dialysis.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Director of PD center, Peking University First Hospital
Other Study IDs: 2022SF38
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Dietary Sodium Intake
Keywords: Dietary Sodium Intake; Peritoneal Dialysis; Equation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop a novel equation for estimating sodium intake in anuric peritoneal dialysis patients, and then to validate its precision and accuracy.

DETAILED DESCRIPTION:
Dietary sodium intake is closely associated with the prognosis of chronic kidney disease (CKD) patients. Previous studies have developed an equation for estimating dietary sodium intake through 24-hour urine sodium in CKD, which are not applicable in peritoneal dialysis patients. This study aims to develop a novel equation for estimating dietary sodium intake in 20 anuric peritoneal dialysis patients, using accurately measured dietary sodium as the dependent variable and peritoneal sodium clearance and its related variables as independent variables, and then to validate the precision and accuracy of the novel equation in another 20 anuric peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis vintage >3 months.
* 18-80 years old.
* No residual renal function (urine volume<200ml/day).
* Continuous ambulatory peritoneal dialysis or manual intermittent peritoneal dialysis.

Exclusion Criteria:

* Peritonitis in the past month.
* Acute systemic infection, cardio-cerebrovascular complications and surgical trauma in the past month.
* Uncorrected hyponatremia (blood sodium<130mmol/L).
* Prescribed with sodium bicarbonate and other drugs containing sodium.
* Prescribed with glucocorticoids and aldosterone antagonists.
* Dysfunction of peritoneal dialysis catheter.
* Malignant tumor receiving radiotherapy and chemotherapy, severe dyspepsia or eating disorder.
* Body fluid loss due to vomit, diarrhea, massive sweating, or other causes.
* Cannot follow the research scheme.
* Refuse to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peritoneal Dialysis Patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
determination coefficient of the novel equation | July 3, 2023, to March 1, 2024
  Determination coefficient will be assessed as the square of the multiple correlation coefficient of the novel equation for estimating sodium intake in peritoneal dialysis.
bias of the novel equation | July 3, 2023, to March 1, 2024
  Bias will be assessed as the median of the difference between the estimated and measured dietary sodium values.
precision of the novel equation | July 3, 2023, to March 1, 2024
  Precision will be assessed as the standard deviation (SD) for the absolute value of difference between the estimated and measured dietary sodium values.
accuracy of the novel equation | July 3, 2023, to March 1, 2024
  Accuracy will be assessed as the percentage of estimates that differed >20% from the measured dietary sodium values (1-P20) .

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, Professor, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No